CLINICAL TRIAL: NCT02285270
Title: A Pilot Study to Investigate Circadian Variations in Brown Adipose Tissue Metabolism in Healthy Volunteers.
Brief Title: Circadian Brown Adipose Tissue Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Daniel Pryma, Primary Investigator, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 819607
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Results first posted 2016-06-17 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: Circadian rhythm; Adipose tissue, brown; Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single group assignment (Other): Diagnostic test/procedure - FDG PET/CT
  Interventions: Device: FDG PET/CT

INTERVENTIONS:
Device: FDG PET/CT — PET/CT is a hybrid imaging modality that allows imaging positron emitting isotopes such as F-18 along with anatomic imaging using x-rays. The physiologic information from the PET component is co-registered with the anatomic information from the CT component, permitting accurate localization and quantification of physiologic processes. The most common clinically used positron emitting radiopharmaceutical is F-18 fluorodeoxyglucose (FDG). It is a glucose analog which is taken up by glucose transporters and phosphorylated to FDG-6P by hexokinase. FDG PET/CT gives a map of relative amount of glucose uptake and phosphorylation over the interval from injection to scan.

SUMMARY:
Brown adipose tissue is poorly understood fat that can metabolize glucose in order to generate heat. Since activated brown fat has a high metabolic rate, it is of great interest as a potential target to combat obesity. However, the signaling and control of brown fat metabolism is poorly understood. Because brown fat uses glucose as its energy source, brown fat metabolism can be imaged with PET/CT using the positron emitting glucose analog F-18 FDG. We have recently shown in mice a striking circadian variation in brown fat metabolism as evidenced by changes in FDG uptake. In this study we endeavor to generate pilot data on a potential circadian variation in brown fat activation in healthy humans.

DETAILED DESCRIPTION:
Brown adipose tissue is a form of fat that is able to metabolize glucose in order to generate heat. When active, it can convert a great deal of glucose into thermal energy. Activation of brown fat could potentially help to combat obesity by increasing the basal metabolic rate. However, activation and signaling of brown fat is poorly understood. In a mouse model, we have recently shown that there is significant circadian variation in brown fat activation and have also discovered the gene that is responsible for the circadian changes (Gerhart-Hines et al, Nature 2013). Specifically, we have shown that in wild type mice, brown fat activation is high at night and low during the day. Whether human brown fat activation has a circadian component is currently unknown. Showing that brown fat activation in humans is subject to similar circadian rhythms as in mice would be an important step in understanding the signaling of activation and may help to elucidate potential strategies to control activation. Positron emission tomography/computed tomography (PET/CT) is a hybrid imaging modality that allows imaging positron emitting isotopes such as fluorine-18 (F-18) along with anatomic imaging using x-rays. The physiologic information from the PET component is co-registered with the anatomic information from the CT component, permitting accurate localization and quantification of physiologic processes. The most common clinically used positron emitting radiopharmaceutical is F-18 fluorodeoxyglucose (FDG). It is a glucose analog which is taken up by glucose transporters and phosphorylated to FDG-6P by hexokinase. However, isomerase, the next enzyme in the glycolytic pathway, is inactive on FDG-6P and so it is largely trapped in the cell. Therefore, FDG PET/CT gives a map of relative amount of glucose uptake and phosphorylation over the interval from injection to scan. Activated brown fat has robust FDG uptake with very intense signal seen. Therefore, FDG PET/CT can be used both to determine whether a person has activated brown fat at the time of the scan as well as to quantify the overall level of metabolism in the fat. Our primary objective is to gather pilot data on the potential presence of circadian variations in brown fat uptake in young, healthy, lean male volunteers. We plan to do this by performing two FDG PET/CT scans 12 hours apart while the patient remains in a temperature and diet controlled environment leading up to both scans. Our primary hypothesis is that brown fat activity will be higher during the day than at night (as human and mouse circadian rhythms are reversed). We will also pair measurement of cortisol with the FDG injections as cortisol levels provide valuable independent information on the circadian rhythm.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and less than 45 years of age
* Able and willing to provide informed consent
* Male gender
* Capable of complying with study procedures and able to lie still in the PET/CT scanner for up to 40 minutes continuously
* Normal fasting glucose (less than 100 mg/dl)
* No evidence of significant concurrent illness
* Follow typical sleep/wake cycle of generally asleep at night and awake during the day

Exclusion Criteria:

* Prior surgery or radiation to the head, neck, or upper chest (except surgeries such as tonsillectomy/adenoidectomy/tympanostomy that would not be expected, in the judgement of the investigator, to have disrupted the adipose tissue in the neck or the upper chest)
* Active addiction or illicit drug abuse
* BMI greater than 25
* Employment in the night shift/3rd shift
* Unable to remain in the Clinical and Translational Research Center (CTRC) for entire 24 hour period.
* Unable or unwilling to maintain peripheral intravenous access for up to 24 hours
* Abnormal liver or kidney function (serum creatinine or transaminase levels greater than 1.5 ULN)
* Subject has any other condition or personal circumstance that, in the judgement of the investigator, might interfere with the collection of complete, high quality data

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pryma, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: The nuclear receptor Rev-erbα controls circadian thermogenic plasticity. — http://www.nature.com/nature/journal/v503/n7476/full/nature12642.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Group Assignment
Started | 10
Completed | 5
Not Completed | 5
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 3
Not completed — Determined to be ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximum Standardized Update Value (SUVmax) in Brown Adipose Tissue FDG Uptake in the Neck or Upper Chest on Evening and Imaging Compared to Morning Imaging
Time Frame: ~12-hours
Population: No patients were analyzed since no patient showed uptake of FDG in brown adipose tissue.
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 0

2. Secondary Outcome: Correlation Between Cortisol Level and Brown Adipose Tissue FDG Uptake
Time Frame: ~12-hours
Population: No patients were analyzed since no patient showed uptake of FDG in brown adipose tissue.
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Total Brown Adipose Tissue FDG Uptake as Measured by Total Volume of Segmented Fat Times the Mean Standardized Uptake Value (SUVmean)
Time Frame: ~12-hours
Population: No patients were analyzed since no patient showed uptake of FDG in brown adipose tissue.
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Arm/Group | Single Group Assignment
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes